CLINICAL TRIAL: NCT00895908
Title: Reducing ADHD by Promoting Social Collaboration and Self-Regulation Skills
Brief Title: Reducing Attention Deficit Hyperactivity Disorder in Kindergarten and Pre-Kindergarten Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karen Bierman, Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34MH085889 (NIH); R34MH085889 (NIH); DDTR B2-MBT
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Psychosocial Intervention; Social Skills Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Comparison of social skill training intervention with active attention control group (academic tutoring)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Friendship Group Intervention (Experimental): Participants will receive the "Friendship Groups" intervention.
  Interventions: Behavioral: Friendship Group
- Individual Tutoring (Active Comparator): Participants will receive individual academic tutoring.
  Interventions: Behavioral: Academic tutoring

INTERVENTIONS:
Behavioral: Friendship Group — Social skills training for 30 sessions, held twice per week over 4 to 5 months
  Arms: Friendship Group Intervention
Behavioral: Academic tutoring — Tutoring to support emergent literacy skills, held 1 to 2 times per week over 4 months
  Arms: Individual Tutoring

SUMMARY:
This study will determine the effectiveness of an intervention for preventing at-risk kindergarten and pre-kindergarten children from developing attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is characterized by inattention, impulsiveness, and hyperactivity. ADHD is not commonly diagnosed until a child has entered formal schooling and shown academic and behavioral adjustment difficulties, but developmental research suggests that risk factors for developing ADHD are evident earlier. A significant number of children start school with high levels of disorganized and inattentive behaviors, which are symptoms of emerging ADHD. This study will test an intervention aimed at preventing the development of ADHD by identifying those at risk for developing ADHD in kindergarten and pre-kindergarten and teaching them self-regulation skills through socialization. These skills have been associated with school success, and they may reduce the likelihood of children developing ADHD.

Participation in this study will last for 4 months, with a follow-up assessment after 1 year. To enroll, child participants will undergo a screening process that will include assessments by their teachers and parents. Eligible child participants will also be assessed by researchers in a classroom setting. They will then be randomly assigned to receive either a play-based intervention, called the Friendship Group, or an individual pre-academic tutoring intervention. Both groups will meet at school. The Friendship Group, which will focus on strengthening attention and self-regulation through social skills, will involve 30 sessions twice a week for 15 weeks. The tutoring intervention, which will focus on strengthening academic skills, will involve one or two sessions a week for 4 months. Participants will be assessed at three time points: pre-intervention, post-intervention, and after 1 year. Assessments will include teacher ratings and direct testing of child attention, language, and pre-academic skills.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or subclinical levels of ADHD symptomatology, based upon teacher and parent report

Exclusion Criteria:

* Presence of sensorimotor disability, frank neurological disorder, or psychosis
* Estimated Full Scale Intelligence Quotient (FSIQ) less than 70
* Very low levels of English proficiency that preclude completion of the assessment battery
* In a temporary custody situation with uncertain outcome

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2013-04-30 (Actual)

PRIMARY OUTCOMES:
Attention deficit hyperactivity disorder (ADHD) symptomatology | Measured pre- and post-treatment and at 12-month follow-up

SECONDARY OUTCOMES:
Social competence | Measured pre- and post-treatment and at 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Bierman, PhD, Principal Investigator — The Pennsylvannia State University

IPD SHARING:
Plan to Share IPD: No